CLINICAL TRIAL: NCT00834223
Title: A Prospective, Multicenter, Open-label, Safety and Preliminary Efficacy Study of the Surgical Implantation of OPKO's Glaucoma Drainage Device (AquashuntTM) in Patients With Refractory Chronic Forms of Open Angle Glaucoma (OAG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Naveed Shams, Opko Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPK-04-101
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Glaucoma
Keywords: refractory chronic forms of open angle glaucoma (OAG); OAG; glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aquashunt (Other): Open label, all subjects receive device.
  Interventions: Device: Aquashunt

INTERVENTIONS:
Device: Aquashunt — A shunt which is implanted into the suprachoroidal space.

SUMMARY:
A prospective, multicenter, open-label, safety and preliminary efficacy study of the surgical implantation of OPKO's glaucoma drainage device (AquashuntTM) in patients with refractory chronic forms of open angle glaucoma (OAG). The primary objective of this study is to evaluate the surgical implantation, safety and preliminary efficacy of the AquashuntTM after implantation in patients with refractory chronic forms of OAG

ELIGIBILITY:
Inclusion Criteria:

Patients of either sex will be eligible for the study if all of the following criteria are met:

1. Patients must be aged 18 years or more.
2. Patients must have a diagnosis of chronic forms of open angle glaucoma in the study eye, which is uncontrolled on maximum tolerated medical treatment with ocular hypotensive medications and has failed glaucoma surgery or is not considered a reasonable candidate for traditional surgery.
3. The patient's documented IOP must be considered by the treating physician to be too high for their glaucoma status.
4. Patients must have BCVA of between 20/400 and Light Perception, or no light perception with pain, in the study eye.
5. Patients must have a BCVA in the fellow eye, which is better than that of the study eye.
6. Patients must be mentally competent and willing to provide informed consent.
7. Patients must be willing to return for all study visits and assessments for at least 3 years after surgery.

Exclusion Criteria

Patients will not be eligible for the study if any of the following criteria are present:

1. Patients with a diagnosis of glaucoma other than open angle glaucoma including active uveitic, active neovascular or recent traumatic glaucoma.
2. Patients with clinically significant corneal disease including corneal dystrophy.
3. Patients with iridocorneal endothelial syndrome.
4. Any previous ocular surgery other than trabeculectomy, trabeculoplasty or cataract surgery and any surgery (including laser) within previous 3 months.
5. Patients with an Anterior Chamber configuration that puts the patient at high risk for the development of angle closure glaucoma.
6. Patients with any recent (within previous 30 days), or current, ocular/periocular inflammation or infection.
7. Patients with a history of extensive keloid formation.
8. Patients who will need ancillary procedures in the study eye at the time of implantation or during the initial one year study period.
9. Patients who have any known intolerance or hypersensitivity to topical anesthetics, mydriatics or components of the device.
10. Patients who are unable to interrupt their anti-coagulant, anti-platelet or NSAID (including aspirin) therapy for at least 3 weeks prior to surgery.
11. Patients who have within the previous 3 months, are currently, or intend to participate in a study with any investigational agent (drug or device).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Primary efficacy measure: The percentage change in IOP from baseline to 6 months and 12 months post-implantation. | 6 and 12 months

SECONDARY OUTCOMES:
Secondary efficacy measure: The change in the number of glaucoma medications from baseline at 6 and 12 months post-implantation. | 6 and 12 months
Safety measures: The incidence of device and procedure-related complications. All adverse events reported, whether deemed related to the treatment or not. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Shams, MD PhD, Study Director — Opko Health
Locations (1):
- Centro Laser, Santo Domingo, Dominican Republic